CLINICAL TRIAL: NCT03310307
Title: Vitamin D3 Treatment Decreases Serum Total Homocysteine Concentrations of Overweight Reproductive Women: Randomized Placebo Controlled Clinical Trail
Brief Title: Vitamin D3 Treatment and Homocysteine Concentrations Among Overweight Reproductive Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Al-Balqa Applied University (Other)
Collaborators: Jordan University of Science and Technology (Other)
Responsible Party: Principal Investigator, Nahla Bayyari, Assistant Professor, Al-Balqa Applied University
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: Hcy-VitD-01
Record Dates: First submitted 2017-10-11; First posted 2017-10-16 (Actual); Last update posted 2017-10-16 (Actual); Status verified 2017-10

CONDITIONS: Homocystinaemia; Vitamin D Deficiency
Keywords: Homocysteine; Overweight; vitamin D3; Reproductive women; RCT
MeSH Terms: conditions — Vitamin D Deficiency; Overweight

STUDY DESIGN:
Masking Description: Double blind
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- vitamin D3 (Active Comparator): 50,000 IU
  Interventions: Drug: Vit D
- Placebo (Placebo Comparator): Similar in size, shape and color to vitamin D3
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Vit D — 50,000 IU
  Other Names: Biodal
  Arms: vitamin D3
Other: Placebo
  Arms: Placebo

SUMMARY:
100 overweight reproductive vitamin D deficient women were divided into two groups; vitamin D (n = 50) and placebo (n = 50). Vitamin D group received treatment dose of 50,000 IU of vitamin D3 per week for 2 consecutive months and placebo group received placebo tablets similar in size, shape and color to vitamin D3 for 2 months also. Total homocysteine concentrations were measured before intervention (basal), on 30 days (one month) and on 60 days (2 months) of intervention. Changes in means of homocysteine concentrations for placebo and vitamin D group over time showed significant difference on 30 and 60 days of intervention. Mean comparisons of homocysteine concentrations and standard error of the means before and after intervention showed statistical significant decrease in homocysteine concentrations among vitamin D group.

ELIGIBILITY:
Inclusion Criteria:

* Overweight (BMI between 25-29.99 kg/m2)
* Had 25(OH)D < 20 ng/mL
* Had normal vitamin B-12 and folic acid levels
* Not diagnosed with any chronic diseases
* Agreed to participat in the study

Exclusion Criteria:

* age < 18 or > 49 years
* BMI > 30 kg/m2 or < 25 kg/m2
* 25 (OH)D level > 20 ng/ml
* tHcy levels greater than 100 µmol/L
* Abnormal vitamin B-12 or folic acid levels
* Chronic diseases
* Pregnant or lactating

Ages: 18 Years to 49 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Attending obstetric and gynecology clinics at King Abdullah University Hospital
Enrollment: 100 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2016-10-30 (Actual)

PRIMARY OUTCOMES:
25(OH)D3 | 2 months
  vitamin D in serum

SECONDARY OUTCOMES:
Homocysteine | 2 months
  serum total homocysteine

CONTACTS AND LOCATIONS:
Overall Officials: Jehan M Hamadneh, FRCOG, Principal Investigator — JUST; Nahla S Al-Bayyari, PhD, Study Chair — BAU
Locations (1):
- King Abdullah University Hospital, Irbid, Jordan

REFERENCES:
- [Derived] Al-Bayyari N, Al-Zeidaneen S, Hailat R, Hamadneh J. Vitamin D3 prevents cardiovascular diseases by lowering serum total homocysteine concentrations in overweight reproductive women: A randomized, placebo-controlled clinical trial. Nutr Res. 2018 Nov;59:65-71. doi: 10.1016/j.nutres.2018.07.012. Epub 2018 Jul 29. PMID 30442234